CLINICAL TRIAL: NCT02080273
Title: The Clinical Investigation of Colgate Total Toothpaste as Compared to Parodontax Toothpaste and Colgate Cavity Protection Toothpaste in Controlling Established Plaque and Gingivitis. (A Six Month Study)
Brief Title: Six Month Plaque and Gingivitis Study Using Colgate Total Toothpaste
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2012-10-CT-BKK-YPZ
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2014-03

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Colgate Cavity Protection toothpaste (Placebo Comparator): Brush whole mouth 2x/day with Colgate Cavity Protection toothpaste. This study treatment is currently marketed/sold in Poland
  Interventions: Drug: Colgate Cavity Protection toothpaste
- Colgate Total toothpaste (Active Comparator): Brush whole mouth 2x/day with Colgate Total toothpaste . This study treatment is currently marketed/sold in Poland
  Interventions: Drug: Colgate Total toothpaste
- Parodontax (Active Comparator): Brush whole mouth 2x/day with Parodontax toothpaste. This study treatment is currently marketed/sold in Poland.
  Interventions: Drug: Parodontax toothpaste

INTERVENTIONS:
Drug: Colgate Cavity Protection toothpaste — 0.76% monofluorophosphate (1000 ppm MFP), Colgate Cavity Protection toothpaste is a control treatment.
  Arms: Colgate Cavity Protection toothpaste
Drug: Colgate Total toothpaste — 0.32% sodium fluoride (1450 ppm NaF) and 0.3% triclosan. Colgate Total toothpaste is the active comparator toothpaste
  Arms: Colgate Total toothpaste
Drug: Parodontax toothpaste — 1400 ppm sodium fluoride (NaF), Parodontax toothpaste is the active comparator toothpaste
  Arms: Parodontax

SUMMARY:
The objective of this randomized, single center, parallel clinical research study is to evaluate the comparative efficacy performance of three dentifrices -Colgate Total Toothpaste, Parodontax Toothpaste and Colgate Cavity Protection Toothpaste in controlling gingivitis and dental plaque in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, ages 18-70, inclusive.
2. Availability for the six-month duration ofthe clinical research study.
3. Good general health.
4. Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
5. Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
6. Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification).
7. Signed Informed Consent Form.

Exclusion Criteria:

1. Presence of orthodontic bands.
2. Presence of partial removable dentures.
3. Tumor(s) of the soft or hard tissues of the oral cavity.
4. Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
5. Five or more carious lesions requiring immediate restorative treatment.
6. Antibiotic use any time during the one month prior to entry into the study.
7. Participation in any other clinical study or test panel within the one month prior to entry into the study.
8. Dental prophylaxis during the past two weeks prior to baseline examinations.
9. History of allergies to oral care/personal care consumer products or their ingredients.
10. On any prescription medicines that might interfere with the study outcome.
11. An existing medical condition which prohibits eating or drinking for periods up to 4 hours.
12. History of alcohol or drug abuse.
13. Pregnant or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terdphong Triratana, Principal Investigator — Mahidol University
Locations (1):
- Mahidol University, Ratchathewi, Bangkok, Thailand

REFERENCES:
- [Derived] Triratana T, Kraivaphan P, Amornchat C, Mateo LR, Morrison BM Jr, Dibart S, Zhang YP. Comparing three toothpastes in controlling plaque and gingivitis: A 6-month clinical study. Am J Dent. 2015 Apr;28(2):68-74. PMID 26087570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment completed by the principal investigator at the clinical site.
Pre-assignment Details: None. There is no wash out/pre-trial period for enrolled subjects. All accepted subjects were randomized upon study enrollment.
Period: Overall Study
Arm/Group | Colgate Cavity Protection Toothpaste | Colgate Total Toothpaste | Parodontax
Started | 45 | 45 | 45
Completed | 45 | 45 | 45
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colgate Cavity Protection Toothpaste | Colgate Total Toothpaste | Parodontax | Total
Number analyzed (Participants) | 45 | 45 | 45 | 135
Age, Continuous [Mean (Full Range); unit: years] | 38.6 [24 to 55] | 38.6 [23 to 54] | 38.4 [21 to 59] | 38.48 [21 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 23 | 69
  Male | 21 | 23 | 22 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 45 | 45 | 45 | 135
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Thailand | 45 | 45 | 45 | 135

OUTCOME MEASURES:

1. Primary Outcome: Dental Plaque Score
Description: Dental Plaque (Quigley-Hein, Turesky Modification Index) Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Colgate Cavity Protection Toothpaste | Colgate Total Toothpaste | Parodontax
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 3.53 (0.37) | 3.55 (0.36) | 3.59 (0.36)
Statistical Analysis 1: Comparison: Colgate Cavity Protection Toothpaste vs Colgate Total Toothpaste vs Parodontax; Means and standard deviations. 1 factor ANOVA to balance treatment groups to show no difference between groups. The null hypothesis states that there is no difference between groups; Test type: Other; p = 0.919, ANOVA

2. Primary Outcome: Dental Plaque Score
Description: as for outcome 1
Time Frame: 3 weeks post treatment use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Colgate Cavity Protection Toothpaste | Colgate Total Toothpaste | Parodontax
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 3.46 (0.15) | 2.98 (0.37) | 3.50 (0.25)
Statistical Analysis 1: Comparison: Colgate Cavity Protection Toothpaste vs Colgate Total Toothpaste vs Parodontax; The null hypothesis states that there is no difference between groups. ANCOVA adjusting for baseline; Test type: Superiority or Other; p = 0.001, ANCOVA — 1 factor ANCOVA to determine difference between groups with baseline as covariate. The F statistic is used to determine significance. If significance is found then a Tukey's multiple comparison is done

3. Primary Outcome: Dental Plaque Score
Description: as for outcome 1
Time Frame: 3 months post treatment use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Colgate Cavity Protection Toothpaste | Colgate Total Toothpaste | Parodontax
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 3.31 (0.42) | 2.45 (0.29) | 3.45 (0.42)
Statistical Analysis 1: Comparison: Colgate Cavity Protection Toothpaste vs Colgate Total Toothpaste vs Parodontax; The null hypothesis states that there is no difference between groups. ANCOVA adjusting for baseline; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

4. Primary Outcome: Dental Plaque Score
Description: as for outcome 1
Time Frame: 6 months post treatment use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Colgate Cavity Protection Toothpaste | Colgate Total Toothpaste | Parodontax
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 3.40 (0.39) | 1.65 (0.45) | 3.23 (0.35)
Statistical Analysis 1: Comparison: Colgate Cavity Protection Toothpaste vs Colgate Total Toothpaste vs Parodontax; The null hypothesis states that there is no difference between groups. ANCOVA adjusting for baseline; Test type: Other; p = 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

5. Primary Outcome: Gingivitis Scores
Description: Gingivitis scale (Loe & Silness Gingival Index) Units on a scale 0 to 3 (0 = no inflammation, 1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Colgate Cavity Protection Toothpaste | Colgate Total Toothpaste | Parodontax
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 1.77 (0.15) | 1.78 (0.20) | 1.77 (0.20)
Statistical Analysis 1: Comparison: Colgate Cavity Protection Toothpaste vs Colgate Total Toothpaste vs Parodontax; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.922, ANOVA

6. Primary Outcome: Gingivitis Scores
Description: as for outcome 5
Time Frame: 3 weeks post treatment use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Colgate Cavity Protection Toothpaste | Colgate Total Toothpaste | Parodontax
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 1.76 (0.17) | 1.65 (0.23) | 1.67 (0.21)
Statistical Analysis 1: Comparison: Colgate Cavity Protection Toothpaste vs Colgate Total Toothpaste vs Parodontax; The null hypothesis states that there is no difference between groups. ANCOVA adjusting for baseline; Test type: Other; p = 0.848, ANCOVA — [p-value comment as in outcome 2, analysis 1]

7. Primary Outcome: Gingivitis Scores
Description: as for outcome 5
Time Frame: 3 months post treatment use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Colgate Cavity Protection Toothpaste | Colgate Total Toothpaste | Parodontax
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 1.63 (0.32) | 1.27 (0.32) | 1.67 (0.34)
Statistical Analysis 1: Comparison: Colgate Cavity Protection Toothpaste vs Colgate Total Toothpaste vs Parodontax; The null hypothesis states that there is no difference between groups. ANCOVA adjusting for baseline; Test type: Other; p = 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

8. Primary Outcome: Gingivitis Scores
Description: as for outcome 5
Time Frame: 6 months post treatment use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Colgate Cavity Protection Toothpaste | Colgate Total Toothpaste | Parodontax
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 1.57 (0.28) | 0.95 (0.26) | 1.47 (0.30)
Statistical Analysis 1: Comparison: Colgate Cavity Protection Toothpaste vs Colgate Total Toothpaste vs Parodontax; The null hypothesis states that there is no difference between groups. ANCOVA adjusting for baseline; Test type: Other; p = 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Colgate Cavity Protection Toothpaste | Colgate Total Toothpaste | Parodontax
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No